CLINICAL TRIAL: NCT04631198
Title: Comparison of the Effects of Conventional Physiotherapy Versus Thoracoabdominal Rebalancing in Reducing Respiratory Complications in Post-operative Patients of Myocardial Revascularization Surgery
Brief Title: Effects of Conventional Physiotherapy and Thoracoabdominal Rebalancing in Post-operative of Myocardial Revascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, KaroliniReis, Principal Investigator, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 5818/20
Record Dates: First submitted 2020-10-19; First posted 2020-11-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Complication
Keywords: Myocardial revascularization surgery; Physical therapy

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized clinical trial. The randomization technique for proposed proposals will be performed using a computer program (www.random.org) containing the coded distribution. The allocation confidentiality will be guaranteed by a randomization list that will be in a remote place, which will prevent the researcher from identifying which intervention will be specified by each patient. The generation of the sequence of numbers will be performed by a researcher "blind" to the study, after selection of the patients by the inclusion criteria. The sequence of numbers one used for randomization will be kept confidential until the exact moment of the beginning of the study. The randomization of the subjects in the proposed groups will be done in two blocks, in which the program will randomly distribute each new participant to one of the blocks: conventional physical therapy group and thoracoabdominal rebalancing group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: GROUP CONTROL (No Intervention): Patients selected for the control group (conventional physiotherapy) will be exposed to respiratory physiotherapy techniques such as vibrocompression, manual passive expiratory therapy, expiratory flow acceleration, fractional inspiration in times, diaphragmatic breaths and aspiration when required
- Active Comparator: INTERVENTION GROUP (Experimental): The patients selected for the intervention group will be submitted to the handling of thoracoabdominal rebalancing as abdominal supports and / or in the ileo-costal space, inspiratory help, scapular waist release, thoracic swing, pectoralis major muscle release and deltoid together with aspiration if necessary.
  Interventions: Other: Thoracoabdominal rebalancing

INTERVENTIONS:
Other: Thoracoabdominal rebalancing — the patients selected for the intervention group will be submitted to the handling of thoracoabdominal rebalancing as abdominal supports and / or in the ileo-costal space, inspiratory help, scapular waist release, thoracic swing, pectoralis major muscle release and deltoid together with aspiration if necessary.
  Arms: Active Comparator: INTERVENTION GROUP

SUMMARY:
When it comes to cardiovascular diseases, surgical or clinical treatment can be cited, and cardiac surgery is considered a complex and large treatment where it involves important organic repercussions that alter the physiological and hemodynamic mechanisms of patients, which can lead to a critical state postoperatively, leading to possible complications that require intensive care at that time. Respiratory complications usually occur frequently in the postoperative period of these surgeries, causing a functional lung capacity to decrease by up to 20%, which may result in atelectasis, pneumonia, pleural effusion, among others. For this reason, physiotherapy usually plays an important role in the treatment of these patients, as it helps to reduce or treat these complications, in addition to promoting motor rehabilitation of patients before myocardial revascularization surgery. For this reason, this study aims to compare the effect of conventional physiotherapy techniques with the management of thoracoabdominal rebalancing in postoperative patients of coronary artery bypass graft. This is a randomized pilot trial in which patients who underwent coronary artery bypass surgery at the Institute of Cardiology of Rio Grande do Sul participate in the study. Patients selected for the control group (conventional physiotherapy) will be exposed to respiratory physiotherapy techniques such as vibrocompression, passive manual expiratory therapy, acceleration of expiratory flow, fractional inspiration in times, diaphragmatic breaths and aspiration when necessary, and patients selected for the intervention group, will appear on the management of thoracoabdominal rebalancing as abdominal supports and / or in the ileo-costal space, inspiratory aid, release of the scapular waist, thoracic swing, release of the pectoralis major and deltoid muscles together with aspiration, if necessary.

DETAILED DESCRIPTION:
Compare the effect of conventional physiotherapy techniques with the management of thoracoabdominal rebalancing in postoperative myocardial revascularization surgery patients. It is a randomized pilot trial in which patients who have undergone myocardial revascularization surgery at the Institute of Cardiology of Rio Grande do Sul will participate in the study.

The study will include individuals over 35 years of age who have myocardial revascularization surgery with prescribed physiotherapeutic treatment, and will be excluded from patients whose patients were intubated and / or remained in mechanics for more than hours or, still, who required non-invasive mechanical norms before or during the collection period.

The work will be submitted to the Research Ethics Committee at the Cardiology Institute of Porto Alegre (CEP-ICFUC). All study participants will receive clear explanations regarding the research, and those who accept to participate in the study voluntarily, will sign the informed consent form, in two copies, one being made available to the participant and the other to researchers. Participants will not be paid, nor will they receive any assistance during or after the end of the survey (466/12).

The benefits of this research will be given in better conducts that prevent or reduce complications and / or respiratory discomfort as well as accelerate the patient's recovery, aiming at hospital discharge more quickly.

Patients selected for the control group (conventional physiotherapy) will be exposed to respiratory physiotherapy techniques such as vibrocompression, passive manual expiratory therapy, acceleration of expiratory flow, fractional inspiration in times, diaphragmatic breaths and aspiration when necessary, and patients selected for the group intervention, will be submitted to the handling of the thoracoabdominal rebalancing as abdominal supports and / or in the ileo-costal space, inspiratory aid, scapular waist release, thoracic swing, release of the pectoralis major and deltoid muscles together with aspiration if any need.

The research presents minimal risk for the participants, which are related to the measurement of variables and / or application of conventional physiotherapy techniques such as vibrocompression, acceleration of expiratory flow, passive manual expiratory therapy that may suggest some discomfort or pain when touching the chest in a sensation of pressure and vibration.

It is expected that patients submitted to the handling of thoracoabdominal rebalancing have lower scores on the pulmonary complications scales, Downes and Raphaelly respiratory discomfort scale and, consequently, show improvement in the other variables.

ELIGIBILITY:
Inclusion Criteria:

* The study will include individuals over 35 years of age who have undergone myocardial revascularization surgery surgery with prescribed physiotherapeutic treatment.

Exclusion Criteria:

* Patients who are intubated and / or remained on mechanical ventilation for more than 48 hours or who needed non-invasive mechanical ventilation before or during the collection period will be excluded.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change in Downes and Raphaelly respiratory distress scale | Immediately before and after 20 minutes
  Points 0-10, where 0 is better and 10 is worse

SECONDARY OUTCOMES:
respiratory rate | Immediately before and after 20 minutes
  irpm
peripheral saturation | Immediately before and after 20 minutes
  SpO2
mean blood pressure | Immediately before and after 20 minutes
  mmHg
Pulmonary auscultation assessment | Immediately before and after 20 minutes
  Wheezing or snoring orstridor
heart rate | Immediately before and after 20 minutes
  bpm

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Eibel, PhD, Study Director — Instituto de Cardiologia
Locations (1):
- Karolini Reis Branco, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hulzebos EH, Van Meeteren NL, De Bie RA, Dagnelie PC, Helders PJ. Prediction of postoperative pulmonary complications on the basis of preoperative risk factors in patients who had undergone coronary artery bypass graft surgery. Phys Ther. 2003 Jan;83(1):8-16. PMID 12495408
- [Background] Cordeiro AM, Souza DC, Quinzani RH, Troster EJ. [Comparison between an upper airway obstruction score and airway endoscopy to detect airway injury associated with endotracheal intubation in children]. J Pediatr (Rio J). 2003 Nov-Dec;79(6):543-9. Portuguese. PMID 14685453
- [Background] Cavenaghi S, Ferreira LL, Marino LH, Lamari NM. Respiratory physiotherapy in the pre and postoperative myocardial revascularization surgery. Rev Bras Cir Cardiovasc. 2011 Jul-Sep;26(3):455-61. doi: 10.5935/1678-9741.20110022. English, Portuguese. PMID 22086584